CLINICAL TRIAL: NCT04634539
Title: IIT2020-02-Gong-GlutaPanc: Phase I Trial of First-line L-glutamine With Gemcitabine and Nab-paclitaxel in Advanced Pancreatic Cancer (GlutaPanc)
Brief Title: Trial of First-line L-glutamine With Gemcitabine and Nab-paclitaxel in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jun Gong, MD (Other)
Collaborators: Emmaus Medical, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Jun Gong, MD, Assistant Professor, Cedars-Sinai Medical Center
Organization: Cedars-Sinai Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT2020-02-Gong-GLUTAPANC
Record Dates: First submitted 2020-11-11; First posted 2020-11-18 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Advanced Pancreatic Adenocarcinoma; Pancreatic Cancer; Pancreatic Ductal Adenocarcinoma
Keywords: gemcitabine; nab-paclitaxel; L-glutamine
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; 130-nm albumin-bound paclitaxel; Glutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gemcitabine + Nab-paclitaxel + L-glutamine (Experimental): For the dose-finding portion of this study, all subjects will receive a combination of L-glutamine, gemcitabine, and nab-paclitaxel which will be preceded by a 1-week (+/- 1 day) administration of L-glutamine. This 1-week administration of L-glutamine will facilitate measurement of baseline and post-glutamine monotherapy plasma metabolite levels prior to addition of gemcitabine and nab-paclitaxel. The combination therapy will be administered over 28-day cycles during the treatment period until disease progression, treatment intolerance, or withdrawal from the study. Patients are expected to be on treatment for 12 cycles.
  Interventions: Drug: Gemcitabine; Drug: Nab-paclitaxel; Drug: L-glutamine

INTERVENTIONS:
Drug: Gemcitabine — Gemcitabine will be administered at 600, 800, or 1000 mg/m2 intravenous (IV) infusion over 30 minutes on days 1, 8, and 15 (every 28-day cycles) during the treatment period. Gemcitabine will be administered immediately after the infusion of nab-paclitaxel. Pre-medication with may be administered per institutional standard practice at the investigator's discretion with gemcitabine.
Drug: Nab-paclitaxel — Nab-paclitaxel will be administered at 75, 100, or 125 mg/m2 intravenous (IV) infusion over 30 minutes on days 1, 8, and 15 (every 28-day cycles) during the treatment period. Nab-paclitaxel will be given first, before infusion of gemcitabine. Pre-medication for nab-paclitaxel may be administered per institutional standard practice at investigator's discretion.
Drug: L-glutamine — The dose levels of L-glutamine in this study will be 0.1, 0.2, and 0.3 g/kg oral twice daily (rounded to nearest 5 g with an upper limit of 15 g twice daily (30 g/day) for any dose level) taken at the same time each day during the treatment period. L-glutamine will be administered for 1 week (+/-1 day) prior to addition of gemcitabine/nab-paclitaxel. Each dose of L-glutamine should be mixed immediately before ingestion with 8 oz. (240 mL) of a cold or room temperature beverage, such as water, milk or apple juice, or 4 oz. (120 mL) to 6 oz. (177 mL) of food such as applesauce or yogurt. L-glutamine is formulated in 5 gram packets as a white crystalline powder in paper-foil-plastic laminate. Complete dissolution is not required prior to administration.
  Other Names: Endari

SUMMARY:
This study will enroll a total of 16 patients with advanced pancreatic cancer at Cedars-Sinai Medical Center. All subjects will receive combination therapy of gemcitabine, nab-paclitaxel, and L-glutamine. The study investigates what the appropriate dosage of L-glutamine is so that there is the lowest risk of side effects, and whether the supplement will make standard chemotherapy of gemcitabine and nab-paclitaxel more effective in treating advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or unresectable, histologically confirmed pancreatic cancer (new diagnosis or recurrent) referred to Cedars-Sinai Medical Center (CSMC), Samuel Oschin Comprehensive Cancer Institute (SOCCI) for first-line chemotherapy. Prior neoadjuvant or adjuvant chemotherapy and/or chemoradiation is allowed but must have been completed >6 months prior to recurrence.
2. Age ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status ≤2 or Karnofsky performance status ≥60%
4. Demonstrate adequate organ and marrow function (within 14 days of study treatment initiation)
5. Have measurable disease based on RECIST 1.1
6. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
7. Female subjects of childbearing potential should be willing to use adequate methods of birth control (hormonal or barrier method of birth control) or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
8. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
9. Willingness to undergo serial peripheral blood draws and provide stool samples during predefined study timepoints and under prespecified conditions (i.e., fasted, morning blood collections).
10. Written informed consent obtained from subject and ability for subject to comply with the requirements of the study.

Exclusion Criteria:

1. Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
2. Has previously received chemotherapy for metastatic disease (treatment with neoadjuvant or adjuvant therapy is allowed so long as progression occurred ≥6 months).
3. Has pre-existing grade ≥3 neuropathy.
4. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
5. Has a known hypersensitivity to any components of the study drugs.
6. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
7. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
8. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
9. Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
10. Has any gastrointestinal disorder (e.g., bowel obstruction) or neurologic condition (e.g., oropharyngeal dysphagia) that may result in impairment of oral intake and/or absorption of study drug in the opinion of the treating investigator.
11. Is currently receiving any parenteral nutrition or enteral (tube) feeding or is planning to use any other nutritional supplement during the study period.
12. Patients on strong CYP2C8 or CYP3A4 inhibitors or inducers within 1 week prior to starting nab-paclitaxel

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-13 (Actual); Primary Completion 2023-07-06 (Actual); Study Completion 2025-06-17 (Actual)

PRIMARY OUTCOMES:
Recommended phase II dose (RP2D) of combination gemcitabine, nab-paclitaxel, and L-glutamine in treatment-naive metastatic pancreatic cancer. | 4 weeks
  The number of dose-limiting toxicities (DLTs), defined as the rate of drug-related grade ≥3 adverse events (AEs) experienced within the first 4 weeks (1 cycle) of study treatment. The RP2D is defined as the dose level closest to the median of the posterior distribution of the maximum tolerated dose (MTD). The MTD is defined as the dose level such that the probability of DLT at the MTD is θ=0.33.

SECONDARY OUTCOMES:
Describe the safety of gemcitabine, nab-paclitaxel and L-glutamine across all investigated dose levels in subjects with untreated advanced pancreatic cancer | From first dose of study treatment until 30 days after the last dose of study treatment (up to approximately 12 months)..
  Number of adverse events as assessed by NCI CTCAE version 5.0
Describe any preliminary evidence of antitumor activity of the combination by assessment of objective response rate as determined by RECIST 1.1 criteria in patients with measurable disease. | From screening/baseline until the last dose of study treatment (up to approximately 12 months).
  Clinical activity of the combination including objective response rate (ORR), defined as proportion of patients with confirmed PR or CR, evaluated every 8 weeks (every 2 cycles ±1 week) according to the revised RECIST guidelines (version 1.1)
Describe any preliminary evidence of antitumor activity of the combination by assessment of progression-free survival as determined by RECIST 1.1 criteria in patients with measurable disease. | From screening/baseline until the last dose of study treatment (up to approximately 12 months).
  Clinical activity of the combination including progression-free survival (PFS), defined as from baseline until date of progression or death due to any cause, evaluated every 8 weeks (every 2 cycles ±1 week) according to the revised RECIST guidelines (version 1.1).
Describe any preliminary evidence of antitumor activity of the combination by assessment of overall survival as determined by RECIST 1.1 criteria in patients with measurable disease. | From screening/baseline until the last dose of study treatment (up to approximately 12 months).
  Clinical activity of the combination including overall survival (OS), defined as from baseline until date of death due to any cause, evaluated every 8 weeks (every 2 cycles ±1 week) according to the revised RECIST guidelines (version 1.1).

CONTACTS AND LOCATIONS:
Overall Officials: Jun Gong, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (2):
- United States (2):
  - Tower Hematology Oncology Medical Group (THO), Beverly Hills, California
  - Cedars-Sinai Medical Center, Los Angeles, California